CLINICAL TRIAL: NCT06262958
Title: REAL-SMART: Recognition and Early Intervention for Alcohol and Substance Abuse in Adolescence, REAL/Systemic Metabolic Alterations Related to Different Psychiatric Disease Categories in Adolescent
Brief Title: Recognition and Early Intervention for Alcohol and Substance Abuse in Adolescence in Adolescent
Acronym: REAL-SMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUH5703459
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Alcoholism; Substance Abuse; Alcohol Dependence; Alcohol-Related Disorders; Substance Use Disorders; Adolescent Behavior; Adolescent Problem Behavior
Keywords: alcohol; substance; abuse; mini-intervention; adolescent
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders; Alcohol-Related Disorders; Adolescent Behavior | interventions — Insemination, Artificial, Heterologous; Therapeutics

STUDY DESIGN:
Intervention Model Description: Clients are randomized into two groups: 1) those receiving TAU and 2) those receiving a mini-intervention for substance and alcohol use an add-on treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (Active Comparator): Clients are receiving normal adolescent psychiatric care, mostly psychotherapy, medications, or both.
  Interventions: Other: Treatment as usual
- e-form of ASSIST alcohol and substance use mini-intervention (Experimental): Clients are receiving normal adolescent psychiatric care, mostly psychotherapy, medications, or both. In addition to that, they will receive a mini-intervention for substance and alcohol use.
  Interventions: Behavioral: ASSIST; Other: Treatment as usual

INTERVENTIONS:
Behavioral: ASSIST — Adolescent psychiatric outpatient will be offered an e-form of ASSIST alcohol and substance use mini-intervention. Results will be compared to those who received TAU.
  Arms: e-form of ASSIST alcohol and substance use mini-intervention
Other: Treatment as usual — Psychotherapy and/or psychotropic drug treatment

SUMMARY:
ASSIST mini-intervention is applied in an electric form in adolescent outpatients to see if it

DETAILED DESCRIPTION:
All 14-20-year-old patients admitted to the Kuopio University Hospital (KUH) adolescent psychiatric outpatient clinic during 2017-2028 are requested to participate. At admission (baseline), the patients are interviewed by the research nurse and asked to fill out questionnaires. The interview includes a semi-structured diagnostic interview (SCID). The participants are interviewed again in six months (follow-up), and the interview is identical to the one conducted in the admission phase.

ELIGIBILITY:
Inclusion Criteria: Admitted to the Kuopio University Hospital (KUH) adolescent psychiatric outpatient clinic during the years 2016-2019

Exclusion Criteria: Unable to understand the questionnaires

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 800 (Estimated)
Dates: Start 2017-08-07 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Decreased consumption of alcohol, tobacco or substances | 6 months
  Decreased scores in ASSIST questionnaire

SECONDARY OUTCOMES:
BDI scores | 6 months
  Decreased scores in BDI questionnaire
GAD scores | 6 months
  Decreased scores in GAD questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tommi T Tolmunen, Docent, Principal Investigator — Professor
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No